CLINICAL TRIAL: NCT00002319
Title: Open Trial of DOX-SL (Stealth Liposomal Doxorubicin Hydrochloride) in the Treatment of Moderate to Severe AIDS-Related Kaposi's Sarcoma
Brief Title: A Study of DOX-SL in the Treatment of AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sequus Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 134C; LTI-30-12
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-01

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Sarcoma, Kaposi; Liposomes; Doxorubicin; Acquired Immunodeficiency Syndrome; Drug Carriers
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Doxorubicin; Liposomes

INTERVENTIONS:
Drug: Doxorubicin hydrochloride (liposomal)

SUMMARY:
To evaluate the safety and effectiveness of Stealth liposomal doxorubicin hydrochloride (DOX-SL) in the long-term treatment of AIDS-related Kaposi's sarcoma (KS) in patients who previously had good responses to DOX-SL in controlled studies of limited duration, or those with KS who discontinued treatment with another Kaposi's sarcoma therapy because of inadequate efficacy or unacceptable toxicity. To provide a defined protocol for Kaposi's sarcoma patients for whom DOX-SL therapy is indicated.

DETAILED DESCRIPTION:
Patients receive DOX-SL every 3 weeks for a maximum of 20 cycles (including any cycles from a previous DOX-SL study). KS lesions are evaluated prior to administration of each treatment, at the end of the final treatment cycle, and at 4 weeks following the end of the final treatment. Patients who respond will be followed every 2 months for up to 1 year. Study treatment may be interrupted for up to 4 months because of complete response, development of opportunistic infections, or adverse drug effects.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylaxis for PCP, cryptococcal, and herpes infections, and antiretroviral therapy provided these doses have been stable for at least 1 month.
* Maintenance therapy for tuberculosis, fungal, and herpes infections.
* Therapy for new episodes of tuberculosis, fungal, and herpes infections except with potentially myelotoxic chemotherapy.
* Foscarnet or ganciclovir for CMV infection.
* Colony stimulating factors and erythropoietin.

Patients must have:

* Moderate to severe AIDS-related Kaposi's sarcoma.
* Documented anti-HIV antibody.
* No active opportunistic infection with mycobacteria, cytomegalovirus, toxoplasma, Pneumocystis carinii, or other microorganisms (if under treatment with myelotoxic drugs).

NOTE:

* Eligible KS patients include those who have discontinued therapy in the control arm of a DOX-SL KS study because of side effects or inadequate efficacy OR other KS patients for whom DOX-SL is believed to be indicated. Patients must not be eligible for other Liposome Technology protocols comparing DOX-SL with established therapies.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Clinically significant cardiac disease.
* Confusion or disorientation.

Concurrent Medication:

Excluded:

* Other cytotoxic cancer chemotherapy.

Patients with the following prior conditions are excluded:

* Prior neoplasms treated with extensive chemotherapy that, in the investigator's opinion, has led to an irreversibly compromised marrow function.
* History of idiosyncratic or allergic reaction to anthracyclines.
* History of major psychiatric illness.

Prior Medication:

Excluded within the past 4 weeks:

* Cytotoxic chemotherapy (other than in a qualifying Liposome Technology protocol).
* Interferon treatment.

Prior Treatment:

Excluded within the past 3 weeks:

* Radiation or electron beam therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - East Bay AIDS Ctr, Berkeley, California
  - Pacific Oaks Med Group, Beverly Hills, California
  - Hematology - Oncology Med Group of San Fernando Valley, Encino, California
  - Dr Becky Miller, Los Angeles, California
  - Apogee Med Group, San Diego, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - UCSF, San Francisco, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Pacific Oaks Med Group, Sherman Oaks, California
  - Dr Mahmoud Mustafa, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - H Lee Moffit Cancer Ctr and Research Institute, Tampa, Florida
  - American Med Research Institute, Atlanta, Georgia
  - Infectious Disease Rsch Consortium of GA / SE Clin Resources, Atlanta, Georgia
  - Northwestern Med Faculty Foundation, Chicago, Illinois
  - Rush Presbyterian Med College, Chicago, Illinois
  - Illinois Masonic Med Ctr / The Cancer Ctr, Chicago, Illinois
  - Henry Ford Hosp, Detroit, Michigan
  - Washington Univ, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - New York Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Graduate Hosp / Tuttleman Cancer Ctr, Philadelphia, Pennsylvania
  - Comprehensive Care Ctr, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Immunological Institute, Houston, Texas
  - Twelve Oaks Hosp, Houston, Texas
  - Virginia Mason Research Center / Clinical Trial Unit, Seattle, Washington

REFERENCES:
- [Background] Jablonowski H, Szelenyi H, Armbrecht C, Mauss S, Niederau C, Strohmeyer G. Liposomal doxorubicin--a new formulation for the treatment of Kaposi's sarcoma: a study on safety and efficacy in AIDS patients. Int Conf AIDS. 1993 Jun 6-11;9(1):397 (abstract no PO-B12-1573)